CLINICAL TRIAL: NCT05078476
Title: Early Active Motion in the Rehabilitation of Flexor Tendon Injuries: Short Splint Versus Relative Motion: a Pilot Randomized Controlled Trial
Brief Title: Rehabilitation of Finger Flexor Tendon Injuries
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021-00929
Record Dates: First submitted 2021-10-13; First posted 2021-10-14 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-06

CONDITIONS: Flexor Tendon Rupture

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manchester Short Splint (Active Comparator): Dorsal splint ending shortly behind the wrist. The splint will be worn for 6 weeks after surgery and the patient will perform active and passive exercises in the splint.
  Interventions: Other: Manchester Short Splint
- Relative Motion Flexion (Experimental): In the relative motion splint the injured finger is positioned in relative flexion in the MCP joint to the adjacent fingers. Additionally to the relative motion flexion splint a wrist orthosis is adapted. Passive and active exercises will be performed out of the splint.
  Interventions: Other: Relative Motion Flexion

INTERVENTIONS:
Other: Manchester Short Splint — 3-5 days after tendon repair the patient will start with hand therapy and the described protocol.
  Arms: Manchester Short Splint
Other: Relative Motion Flexion — 3-5 days after tendon repair the patient will start with hand therapy and the described protocol.
  Arms: Relative Motion Flexion

SUMMARY:
The primary objective is to compare the two different rehabilitation protocols relative motion flexion and short splint regarding patients'satisfaction in patients with flexor tendon injuries in Zone I and II after 13 and 26 weeks post-surgery.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent as documented by signature
* ≥ 18 years old
* Understanding of the German language (written and oral)
* Single and multiple finger injuries
* Primary flexor tendon injuries in Zone I-V for the fingers and/ or thumb
* Treated by the hand surgery department at the Inselspital Bern
* Treated with at least a 4-strand core suture

Exclusion Criteria:

* < 18 years old
* Inability to follow the procedures of the study, e.g. due to language problems, diagnosed psychological disorders or dementia of the patients
* Replantation of the injured finger
* Fracture of the injured finger
* Primary tendon reconstructions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in patient satisfaction | 13 and 26 weeks after tendon repair
  The satisfaction with the outcome will be evaluated by asking the patient a Single Assessment Numeric Evaluation (SANE) question: "How satisfied are you with your hand on a scale from 0 (not satisfied at all) to 10 (fully satisfied)?

SECONDARY OUTCOMES:
Michigan Hand Questionnaire (MHQ) | 6, 13 and 26 weeks after tendon repair
  The MHQ is a hand specific questionnaire used to measure the ability in daily function. The total score ranges from 0 to 100, with higher scores indicating better performance.
Disabilities of Shoulder, Arm and Hand Questionnaire | 6, 13 and 26 weeks after tendon repair
  The DASH questionnaire is a region-specific outcome instrument. The patient will rate 30-items about disability or symptoms by rating the degree of difficulty in doing various activities. The scores of all items are used to calculate a score ranging from 0 (no disability) to 100 (most severe disability).
Range of motion | 6, 13 and 26 weeks after tendon repair
  The range of motion will be measured with a goniometry.
Grip Strength | 13 and 26 weeks after tendon repair
  Grip Strength will be measured with the JAMAR Dynamometer.
Level of pain | 6, 13 and 26 weeks after tendon repair
  The patient will be asked to rate the pain from 0 to 10. 0 indicates no pain, 10 the worst possible pain. The patient rate the pain while relaxed and during exercises.
Number of therapy sessions | 26 weeks after tendon repair
  The number of therapy sessions will be counted after 26 weeks or at the end of of therapy if after 26 weeks measurement.
Ten Test | 6, 13 and 26 weeks after tendon repair
  The Ten Test is a measure of discriminative sensation, whereby the patient describes the sensation from no sensation "0" to normal sensation "10" on an 11-point Likert scale.
Patients specific function scale | 6, 13 and 26 weeks after tendon repair
  The patient defines three to five activities that are difficult or that he/she is unable to perform due to the hand injury. The patient is asked to rate the difficulty associated with each activity from 0 to 10. 0 is defined as not able to do the activity and 10 is able to do the activity normally.
Work Productivity and Activity Impairment Questionnaire | 6, 13 and 26 weeks after tendon repair
  The WPAI is a quantitative assessment of absenteeism, presenteeism, and overall productivity loss attributable to a specific health problem during the previous 7 days.
Rupture rate/ Complications | 26 weeks after tendon repair
  Tendon rupture will be documented
Complications | 26 weeks after tendon repair
  complications will be documented (e.g. CRPS, infection)

CONTACTS AND LOCATIONS:
Overall Officials: Bernadette Tobler, Dr. phil., Principal Investigator — Inselspital, Bern Universtiy Hospital
Locations (1):
- Inselspital, Bern University Hospital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hardy M, Feehan L, Savvides G, Wong J. How controlled motion alters the biophysical properties of musculoskeletal tissue architecture. J Hand Ther. 2023 Apr-Jun;36(2):269-279. doi: 10.1016/j.jht.2022.12.003. Epub 2023 Apr 5. PMID 37029054